CLINICAL TRIAL: NCT03112720
Title: A Comparison of the Efficacy of Sphenopalatine Ganglion (SPG) Block With 5% Lidocaine Versus Epidural Blood Patch (EBP) for the Treatment of Post-Dural Puncture Headache (PDPH)
Brief Title: Therapeutic Epidural Patch Versus Pain Block in the Midface for Headache
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: no enrollment after covid pandemic
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: New Jersey Medical School (Other)
Responsible Party: Principal Investigator, William Grubb, M.D., Clinical Associate Professor, Anesthesia, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro20140000026
Record Dates: First submitted 2014-09-03; First posted 2017-04-13 (Actual); Results first posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Postdural Puncture Headache
MeSH Terms: conditions — Post-Dural Puncture Headache | interventions — Blood Patch, Epidural; Sphenopalatine Ganglion Block

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Epidural blood patch (Active Comparator): 20ml of sterile blood is obtained from the patients arm and placed in the epidural space using standard sterile epidural access.
  Interventions: Device: Epidural Blood Patch
- Sphenopalatine Ganglion Block (Experimental): Cotton tip applicators are used to deliver lidocaine to the posterior nares in the area of skin overlying the Sphenopalatine gangion
  Interventions: Drug: Sphenopalatine Ganglion Block

INTERVENTIONS:
Device: Epidural Blood Patch — A device: 17 gauge Tuohy needle will be placed to the epidural space using the loss of resistance technique. Once positioned a sterile stylet will be replaced within the needle to maintain the sterility of the epidural space. A tourniquet may be used to identify a peripheral venous site, which will be sterilely prepped with betadine x3 and then chloraprep. Venipuncture will be performed with a device: 20gauge or larger needle. 20mL of blood will be aspirated in a sterile system into an appropriately sized syringe. After sterile transfer, this autologous blood will be slowly injected into the epidural space.
  Arms: Epidural blood patch
Drug: Sphenopalatine Ganglion Block — The drug: 5% lidocaine ointment, a local anesthetic, will be applied to the end of a device: long channeled cotton tipped applicator inserted into both nares and placed over the mucosa in the area of posterior aspect of the middle ethmoid, toward the presumed anatomic location of the sphenopalatine ganglion, evidenced by a slight resistance at the appropriate depth. 5mL of drug: 1% lidocaine solution will then be injected into the hollow shaft of the device: applicator and allowed to topically anesthetize the ganglion by gravity flow for 30 minutes.
  Arms: Sphenopalatine Ganglion Block

SUMMARY:
The purpose of this study is to compare a pain block in the midface, versus the traditional, more invasive, therapeutic epidural patch for the treatment of headaches

DETAILED DESCRIPTION:
The sphenopalatine nerve block has been used to treat headaches. Patients have headaches after epidural access from post dural puncture. We need to know if sphenopalatine nerve block will help the patient with the headache.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ages 13-92
* Subjects have medical diagnosis of PDPH and require treatment
* Subjects who signed consent/assent

Exclusion Criteria:

* <13 years of age
* Pregnancy
* Subjects with heart failure
* Subjects already being treated with lidocaine patch or other vehicle for chronic pain
* Non-english speaking subjects
* Subjects with platelets <100,000
* Subjects that are septic
* Subjects with an allergy to lidocaine
* Subjects with known nasal polyps
* Subjects with recent neurological event
* Subjects on anticoagulant therapy
* Subjects that received prior therapy with SPG block or EBP

Ages: 13 Years to 92 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-09; Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Grubb, DDS, MD, Principal Investigator — Rutgers Robert Wood Johnson Medical School
Locations (2):
- United States (2):
  - New Jersey Pain Center, New Brunswick, New Jersey
  - RWJUH/Barnabus, New Brunswick, New Jersey

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Epidural Blood Patch Group: 20ml of sterile blood is obtained from the patients arm and placed in the epidural space using standard sterile epidural access.
  Epidural Blood Patch: A device: 17 gauge Tuohy needle will be placed to the epidural space using the loss of resistance technique. Once positioned a sterile stylet will be replaced within the needle to maintain the sterility of the epidural space. A tourniquet may be used to identify a peripheral venous site, which will be sterilely prepped with betadine x3 and then chloraprep. Venipuncture will be performed with a device: 20gauge or larger needle. 20mL of blood will be aspirated in a sterile system into an appropriately sized syringe. After sterile transfer, this autologous blood will be slowly injected into the epidural space.
- Sphenopalatine Ganglion Block Group: Cotton tip applicators are used to deliver lidocaine to the posterior nares in the area of skin overlying the Sphenopalatine gangion
  Sphenopalatine Ganglion Block: The drug: 5% lidocaine ointment, a local anesthetic, will be applied to the end of a device: long channeled cotton tipped applicator inserted into both nares and placed over the mucosa in the area of posterior aspect of the middle ethmoid, toward the presumed anatomic location of the sphenopalatine ganglion, evidenced by a slight resistance at the appropriate depth. 5mL of drug: 1% lidocaine solution will then be injected into the hollow shaft of the device: applicator and allowed to topically anesthetize the ganglion by gravity flow for 30 minutes.
Period: Overall Study
Arm/Group | Epidural Blood Patch Group | Sphenopalatine Ganglion Block Group
Started | 5 | 3
Completed | 5 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Epidural Blood Patch | Sphenopalatine Ganglion Block | Total
Number analyzed (Participants) | 5 | 3 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 3 | 8
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 30.4 [27 to 33] | 24.3 [23 to 34] | 29.25 [23 to 34]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Headaches With a VAS Score >8/10 Prior to Initiation of Either Therapy
Description: Outcome measure will entail recording patient self-reported pain scores to quantify the level of headache pain using the Visual analog scale, meaning 0 - No pain, 1-3 - Mild Pain, 4-6 - Moderate Pain, 7-10 - Severe Pain, by way of in person assessment by pain questionnaire just prior to initiation of either therapy (Epidural blood patch vs Sphenopalatine Ganglion Block).
Time Frame: Prior to initiation of therapy (Epidural blood patch vs Sphenopalatine Ganglion Block).
Population: patients having known dural puncture after epidural access for analgesia
Measure: Number; unit: headache with VAS >8/10
Arm/Group | Epidural Blood Patch Group | Sphenopalatine Ganglion Block Group
Number analyzed (Participants) | 5 | 3
headache with VAS >8/10 | 1 | 1

2. Primary Outcome: Number of Participants With a Headache Vas 8/10 at 30 Minutes Following Either Therapy.
Description: Self-reported pain scores to quantify the level of headache pain using the Visual analog scale (as defined within the description of outcome 1 above) by way of in person assessment by pain questionnaire at 30 minutes following either therapy (Epidural blood patch vs Sphenopalatine Ganglion Block).
Time Frame: At 30 minutes following either therapy.
Population: patients having a known dural puncture associated with epidural placement for analgesia
Measure: Count of Participants; unit: Participants
Arm/Group | Epidural Blood Patch Group | Sphenopalatine Ganglion Block Group
Number analyzed (Participants) | 5 | 3
Participants | 1 | 1

3. Primary Outcome: Number of Participants With a Headache Vas 8/10 at 60 Minutes Following Either Therapy.
Description: Self-reported pain scores to quantify the level of headache pain using the Visual analog scale (as defined within the description of outcome 1 above) by way of in person assessment by pain questionnaire at 60 minutes following either therapy (Epidural blood patch vs Sphenopalatine Ganglion Block).
Time Frame: At 60 minutes following either therapy.
Population: patients with headache after known dural puncture after epidural access for analgesia
Measure: Count of Participants; unit: Participants
Arm/Group | Epidural Blood Patch Group | Sphenopalatine Ganglion Block Group
Number analyzed (Participants) | 5 | 3
Participants | 1 | 0
Statistical Analysis 1: Comparison: Epidural Blood Patch Group vs Sphenopalatine Ganglion Block Group; Test type: Other; p < 0.01, Chi-squared; Odds Ratio (OR) = 1.5; < 0.01 study terminated because of covid and no meaningfull numbers participated

ADVERSE EVENTS:
Time Frame: 48 hours
Arm/Group | Epidural Blood Patch Group | Sphenopalatine Ganglion Block Group
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/3
Other Adverse Events (participants affected / at risk) | 0/5 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-05): https://cdn.clinicaltrials.gov/large-docs/20/NCT03112720/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-13): https://cdn.clinicaltrials.gov/large-docs/20/NCT03112720/ICF_001.pdf